CLINICAL TRIAL: NCT04985409
Title: Stepping Up: A Trial of Activity Monitoring Devices in Patients Undergoing Autologous Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Paquette, Medical Director, Blood and Marrow Transplant Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CSHS0523
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma; Lymphoma; Transplant-Related Disorder
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects who are randomized to not get feedback about their activity will not be aware that there is another group that is receiving feedback
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback (Experimental): Participants in the intervention arm will receive a Fitbit upon admission and will receive feedback from the activity tracker and the in-room TV screen as demonstrated by the Study Navigator. Study participants in this arm will be engaging with their physicians around achievement of daily step goals by viewing the in-room TV display of their daily step counts on rounds.
  Interventions: Behavioral: Feedback
- Control (No Intervention): Subjects in the control arm will receive a Fitbit upon admission for their transplant but neither the physician, nurse, nor patient will receive any feedback from the device. They will be blinded to any data capture by their activity monitor. Nurses and doctors will not monitor ambulation with the activity monitor, they will use standard methods to encourage ambulation.

INTERVENTIONS:
Behavioral: Feedback — The system uses Sonifi health (TV content and visualizations) and Fitabase (3rd party server to process Fitbit data and export to Sonifi). The system utilizes the patient's TVs to engage the patient and multidisciplinary team in monitoring ambulation status.
  Arms: Feedback

SUMMARY:
The purpose the research is to obtain preliminary data about the change in fitness from admission to discharge in patients undergoing an Autologous Stem Cell Transplant (ASCT) , assessed by the 6 minute walk test as the primary objective and the SF-36 as the secondary objective. All subjects will wear a Fitbit monitor while admitted for the ASCT to record their daily activity.

DETAILED DESCRIPTION:
This study will enroll 20 subjects with a diagnosis of multiple myeloma or lymphoma (10 with each diagnosis) scheduled to undergo ASCT at Cedars-Sinai Medical Center.

After signing the informed consent form, intake data will be collected on all subjects will include age, diagnosis, Karnofsky performance status, and comorbidity index. Subjects will complete an SF-36 questionnaire that assesses their functional and emotional status. Each subject will undergo a 6-minute walk test (6MWT) while wearing a Fitbit monitor to record the number of steps taken. After admission, subjects will be randomly assigned to either the control or intervention group. Subjects in the control arm will receive an activity monitor but the physician, nurse, and patient will not receive any feedback from the device. Patients will be blinded to any data capture from their activity monitor. Participants in the intervention arm will receive an activity monitor and they will receive feedback from the activity tracker and the in-room TV screen. Study participants in this arm will engage with their physicians and nurses around achievement of daily step goals by viewing the in-room TV display of daily step counts on rounds. After discharge, all subjects will again complete the SF-36 questionnaire and perform a 6MWT at a routine clinic visit, within 30 days of the transplant procedure. Descriptive statistics in the form of mean and standard deviation will be used to summarize patient physical activity as measured by 6MWT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple myeloma or lymphoma with plan to undergo autologous stem cell transplant
* at least 18 years of age
* English or Spanish speaking
* have access to an IOS or Android device
* able to provide informed consent.

Exclusion Criteria:

* pre-existing physical limitations which would preclude achievement of the ambulation goals
* inability to wear the activity monitor
* Jehovah's Witness patients enrolled in the bloodless transplant program are excluded as they require strict bed rest for long periods of time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Fitness measured by 6 minute walk test after discharge | 3-4 weeks
  Standard 6 minute walk test will be performed

SECONDARY OUTCOMES:
Fitness assessed by SF-36 questionnaire after discharge | 3-4 weeks
  Standard SF-36 questionnaire will be completed

CONTACTS AND LOCATIONS:
Overall Officials: Ron Paquette, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No